CLINICAL TRIAL: NCT00002370
Title: Pharmacokinetics Study of Intravenous Itraconazole Followed by Oral Dosing at 200 Mg Twice Daily in Patients With Advanced HIV Infection
Brief Title: Study of Itraconazole in Patients With Advanced HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janssen, LP (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 254B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: HIV Infections
Keywords: Itraconazole; Administration, Oral; Antifungal Agents; Acquired Immunodeficiency Syndrome; Drug Administration Schedule
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Itraconazole

INTERVENTIONS:
Drug: Itraconazole

SUMMARY:
To demonstrate a dosage regimen for intravenous itraconazole that produces a plasma concentration range comparable to that obtained after currently used oral dosages of itraconazole oral solution; and to obtain preliminary safety data in patients with advanced HIV disease.

DETAILED DESCRIPTION:
Patients will receive intravenous itraconazole solution twice daily for 2 days and then once daily for five additional days. Patients then randomized to receive twice-daily or once-daily itraconazole oral solution for an additional 28 days.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Antiretroviral therapy providing patient has already been on a stable, unchanged regimen for 8 weeks prior to study entry.

Patients must have:

* Documented HIV infection.
* CD4 lymphocyte count < 300 cells/mm3.
* No clinically significant abnormalities, elicited by history and physical examination.
* No clinically significant abnormalities in blood count, biochemical profile, or urinalysis within 2 weeks of study entry.
* Negative urine screening.
* No clinically significant abnormalities of electrocardiogram.

Prior Medication:

Allowed:

Antiretroviral therapy providing patient has been on a stable, unchanged regimen for 8 weeks prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Acute opportunistic infection or other significant concurrent illness that would preclude participation for the required 36 days.
* Unable to swallow oral solution.
* Obesity greater than 25% of ideal body weight.

Concurrent Medication:

Excluded:

* Rifampin.
* Rifabutin.
* Phenobarbital.
* Phenytoin.
* Carbamazepine.
* Digoxin.
* Warfarin.
* Midazolam.
* Triazolam.
* Terfenadine.
* Astemizole.
* Cisapride.
* H2 blockers.
* Omeprazole.
* Continual antacids.
* Didanosine.
* Any medication known to affect absorption, metabolism or excretion of imidazole or azole compounds.

Patients with the following prior symptoms and conditions are excluded:

* Previous hypersensitivity to azole antifungals.
* History of surgical procedure that may interfere with absorption of itraconazole.
* History of significant blood loss in the previous 30 days.

Prior Medication:

Excluded:

Excluded within 15 days prior to study entry:

* Rifampin.
* Rifabutin.
* Phenobarbital.
* Phenytoin.
* Carbamazepine.
* Digoxin.
* Warfarin.
* Midazolam.
* Triazolam.

Excluded within 8 weeks prior to study entry:

* Change in antiretroviral therapy.

Risk Behavior:

Excluded:

Patients who chew tobacco or regularly smoke more than 10 cigarettes per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36

CONTACTS AND LOCATIONS:
Locations (1):
- Erie County Med Ctr / Pharmacy D, Buffalo, New York, United States